CLINICAL TRIAL: NCT03960775
Title: The Influence of Perioperative Administration of Dexmedetomidine on Inflammation Response and Postoperative Recovery in Patients Undergoing Robot or Laparoscopic Assisted Gastrectomy; Double Blind Randomized Controlled Trial
Brief Title: The Influence of Perioperative Administration of Dexmedetomidine on Inflammation Response and Postoperative Recovery in Patients Undergoing Robot or Laparoscopic Assisted Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2019-0055
Record Dates: First submitted 2019-04-29; First posted 2019-05-23 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Gastric Cancer; Gastrostomy
Keywords: gastric cancer; laparoscopic gastrectomy; robotic gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Investigator prepared the drug and participant and outcomes assessor were blind to the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (dexmedetomidine) (Experimental): dexmedetomidine infusion group
  Interventions: Drug: dexmedetomidine
- Group B (saline) (Placebo Comparator): normal saline infusion group
  Interventions: Drug: saline

INTERVENTIONS:
Drug: dexmedetomidine — Dexmedetomidine infusion (0.4㎍/kg/hr) from anesthetic induction until the start of closure of peritoneum.
  Arms: Group A (dexmedetomidine)
Drug: saline — Saline infusion during same time period.
  Arms: Group B (saline)

SUMMARY:
Many studies have shown that inflammation has an important effect on the development, progression, and also response to treatment of tumors. Dexmedetomidine is a potent and selective alpha 2 receptor agonist, known to have a sedative, analgesic and immune-controlling effect. The purpose of this study is to investigate the effect of dexmedetomidine during surgery on postoperative inflammatory response and surgical recovery in gastric cancer patients undergoing robot or laparoscopic gastrectomy.

DETAILED DESCRIPTION:
* Experimental group (Dexmedetomidine group) Continuous IV Precedex™ using infusion pump (Terufusion TE-311, Terumo, Tokyo, Japan) during surgery (from immediately after induction to before starting peritoneum closure) Infusion rate 0.4μg/kg/hr
* Control group (normal saline group) Continuous IV normal saline using infusion pump (Terufusion TE-311, Terumo, Tokyo, Japan) during surgery Infusion rate 0.4μg/kg/hr

ELIGIBILITY:
Inclusion Criteria:

* 1. 20-70 yrs old patients
* 2. Scheduled for robot or laparoscopic gastrectomy
* 3. Body weight under 90kg and BMI under 32

Exclusion Criteria:

* 1. Emergency operation
* 2. Reoperation
* 3. Co-operation with other surgery department
* 4. Co-operation with other organs (except cholecystectomy)
* 5. Patients with history of heart failure (unstable angina, congestive heart failure)
* 6. Patients with history of arrhythmia (specially AV nodal block), ventricular conduction problem
* 7. Patients with history of uncontrolled hypertension (diastolic BP >110mmHg), extremely bradycardia (HR <45 bpm on ECG)
* 8. Patients with history of cerebrovascular disease (cerebral hemorrhage, cerebral ischemia
* 9. Patients who is steroid user
* 10. Patients who is beta blocker user
* 11. Patients with history of liver failure, renal failure, allergic to medicine
* 12. Patients with history of uncontrolled psychiatric disease (PTSD, anxiety, depression)
* 13. Patients who cannot read the consent form (examples: Illiterate, foreigner)
* 14. Patients who withdraw the consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
CRP level in blood | Preoperative outpatient 1 day visit
  To evaluate the effect of dexmedetomidine on the level of CRP in patients undergoing robot or laparoscopic gastrectomy, CRP level was measured 5 times above time points.
CRP level in blood | Immediately after surgery
  To evaluate the effect of dexmedetomidine on the level of CRP in patients undergoing robot or laparoscopic gastrectomy, CRP level was measured 5 times above time points.
CRP level in blood | POD 1 day
  To evaluate the effect of dexmedetomidine on the level of CRP in patients undergoing robot or laparoscopic gastrectomy, CRP level was measured 5 times above time points.
CRP level in blood | POD 2 day
  To evaluate the effect of dexmedetomidine on the level of CRP in patients undergoing robot or laparoscopic gastrectomy, CRP level was measured 5 times above time points.
CRP level in blood | POD 3 day
  To evaluate the effect of dexmedetomidine on the level of CRP in patients undergoing robot or laparoscopic gastrectomy, CRP level was measured 5 times above time points.
CRP level in blood | discharge day (Postoperative day 5)
  To evaluate the effect of dexmedetomidine on the level of CRP in patients undergoing robot or laparoscopic gastrectomy, CRP level was measured 5 times above time points.
CRP level in blood | first visit after surgery (POD 1 month)
  To evaluate the effect of dexmedetomidine on the level of CRP in patients undergoing robot or laparoscopic gastrectomy, CRP level was measured 5 times above time points.

SECONDARY OUTCOMES:
cytokine (IFN-r, TNF-a, IL-6, IL-8, IL-10, HMGB1) level | Baseline (Preoperative outpatient visit)
  To evaluate the effect of dexmedetomidine on the level of cytokine in patients undergoing robot or laparoscopic gastrectomy, cytokine level was measured 7 times above time points using ELISA analysis.
cytokine (IFN-r, TNF-a, IL-6, IL-8, IL-10, HMGB1) level | immediately after surgery (POD 0)
  To evaluate the effect of dexmedetomidine on the level of cytokine in patients undergoing robot or laparoscopic gastrectomy, cytokine level was measured 7 times above time points using ELISA analysis.
cytokine (IFN-r, TNF-a, IL-6, IL-8, IL-10, HMGB1) level | POD 1 day
  To evaluate the effect of dexmedetomidine on the level of cytokine in patients undergoing robot or laparoscopic gastrectomy, cytokine level was measured 7 times above time points using ELISA analysis.
cytokine (IFN-r, TNF-a, IL-6, IL-8, IL-10, HMGB1) level | POD 2 day
  To evaluate the effect of dexmedetomidine on the level of cytokine in patients undergoing robot or laparoscopic gastrectomy, cytokine level was measured 7 times above time points using ELISA analysis.
cytokine (IFN-r, TNF-a, IL-6, IL-8, IL-10, HMGB1) level | POD 3 day
  To evaluate the effect of dexmedetomidine on the level of cytokine in patients undergoing robot or laparoscopic gastrectomy, cytokine level was measured 7 times above time points using ELISA analysis.
cytokine (IFN-r, TNF-a, IL-6, IL-8, IL-10, HMGB1) level | discharge day (Postoperative day 5)
  To evaluate the effect of dexmedetomidine on the level of cytokine in patients undergoing robot or laparoscopic gastrectomy, cytokine level was measured 7 times above time points using ELISA analysis.
cytokine (IFN-r, TNF-a, IL-6, IL-8, IL-10, HMGB1) level | first visit after surgery (POD 1 month)
  To evaluate the effect of dexmedetomidine on the level of cytokine in patients undergoing robot or laparoscopic gastrectomy, cytokine level was measured 7 times above time points using ELISA analysis.
WBC level | Baseline (Preoperative outpatient visit)
  To evaluate the effect of dexmedetomidine on the level of WBC in patients undergoing robot or laparoscopic gastrectomy, WBC level was measured 7 times above time points.
WBC level | immediately after surgery (POD 0)
  To evaluate the effect of dexmedetomidine on the level of WBC in patients undergoing robot or laparoscopic gastrectomy, WBC level was measured 7 times above time points.
WBC level | POD 1 day
  To evaluate the effect of dexmedetomidine on the level of WBC in patients undergoing robot or laparoscopic gastrectomy, WBC level was measured 7 times above time points.
WBC level | POD 2 day
  To evaluate the effect of dexmedetomidine on the level of WBC in patients undergoing robot or laparoscopic gastrectomy, WBC level was measured 7 times above time points.
WBC level | POD 3 day
  To evaluate the effect of dexmedetomidine on the level of WBC in patients undergoing robot or laparoscopic gastrectomy, WBC level was measured 7 times above time points.
WBC level | discharge day (Postoperative day 5)
  To evaluate the effect of dexmedetomidine on the level of WBC in patients undergoing robot or laparoscopic gastrectomy, WBC level was measured 7 times above time points.
WBC level | first visit after surgery (POD 1 month)
  To evaluate the effect of dexmedetomidine on the level of WBC in patients undergoing robot or laparoscopic gastrectomy, WBC level was measured 7 times above time points.
postoperative pain score (NRS 0~10) | postoperative 0~2hours
  To evaluate the effect of dexmedetomidine on score of postoperative pain in patients undergoing robot or laparoscopic gastrectomy, NRS was measured during postoperative 48 hours.
postoperative pain score (NRS 0~10) | 2~4 hours
  To evaluate the effect of dexmedetomidine on score of postoperative pain in patients undergoing robot or laparoscopic gastrectomy, NRS was measured during postoperative 48 hours.
postoperative pain score (NRS 0~10) | 4~8 hours
  To evaluate the effect of dexmedetomidine on score of postoperative pain in patients undergoing robot or laparoscopic gastrectomy, NRS was measured during postoperative 48 hours.
postoperative pain score (NRS 0~10) | 8~12 hours
  To evaluate the effect of dexmedetomidine on score of postoperative pain in patients undergoing robot or laparoscopic gastrectomy, NRS was measured during postoperative 48 hours.
postoperative pain score (NRS 0~10) | 12~24 hours
  To evaluate the effect of dexmedetomidine on score of postoperative pain in patients undergoing robot or laparoscopic gastrectomy, NRS was measured during postoperative 48 hours.
postoperative pain score (NRS 0~10) | 24~48 hours
  To evaluate the effect of dexmedetomidine on score of postoperative pain in patients undergoing robot or laparoscopic gastrectomy, NRS was measured during postoperative 48 hours.
postoperative any unwanted admission | postoperative 1 month
  To evaluate the effect of dexmedetomidine on postoperative any unwanted admission in patients undergoing robot or laparoscopic gastrectomy, postoperative any unwanted admission was checked during postoperative 1 month.
gas passing out time | gas passing time immediately after surgery
  To evaluate the effect of dexmedetomidine on gas passing in patients undergoing robot or laparoscopic gastrectomy, gas passing out time was checked.
HOD (hospital days) | total days from operation to discharge up to 2 weeks
  To evaluate the effect of dexmedetomidine on hospital day (HOD) in patients undergoing robot or laparoscopic gastrectomy, discharge day was checked.

CONTACTS AND LOCATIONS:
Overall Officials: Na Young Kim, MD, Principal Investigator — Severance Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea